CLINICAL TRIAL: NCT04742504
Title: Interaction Between Benralizumab and Basophils in Eosinophilic Asthma. Discovering a New Role of an Old Asthma Player: BASEAS STUDY (Basophils in Eosinophilic Asthma)
Brief Title: Interaction Between Benralizumab and Basophils in Eosinophilic Asthma
Acronym: BASEAS
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: ESR-20-20764
Record Dates: First submitted 2021-01-07; First posted 2021-02-08 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Asthma; Eosinophilic
Keywords: Asthma; Basophils; anti-receptor de interleukin 5; microRNAs; Benralizumab
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — benralizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, sputum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BENRA Treated Patients: Patients with severe eosinophilic asthma who will be treated with benralizumab (Fasenra®, Astra Zeneca) will be able to participate in a volunteer manner in the study after sing informed consent.
  Interventions: Biological: BENRALIZUMAB
- Non BENRA TREATED PATIENTSP: patients with controlled severe asthma requiring high-dose inhaled corticosteroids plus long-acting beta agonists (with or without oral corticosteroids) but without request of benralizumab (Fasenra®, Astra Zeneca) treatment will be recruited

INTERVENTIONS:
Biological: BENRALIZUMAB — The decision of the patients treatment with benralizumab (Fasenra®, Astra Zeneca) included in the study will not come in any case influenced by their participation in the study but will be made in accordance with the clinical criteria established by the Asthma Multidisciplinary Unit (UMA).
  Groups: BENRA Treated Patients

SUMMARY:
In this study, investigators want to evaluation of the impact of benralizumab (Fasenra®, Astra Zeneca) on different cell populations, including basophils and innate lymphoid cells, and several biomarkers, such as miRNAs, cadena α dek receptor pra la interleukin % (IL5Rα) and soluble IL5Rα in patients with severe eosinophilic asthma. For this, basophil and innate cells type 2 (ILC2) populations will be monitored in different point-time of treatment: 8 week (V1), 6 months (V2) and 1 year (V3) in blood and sputum samples. Also, follow-up IL5Rα expression on a cell surface of eosinophils, basophils and ILC2 from peripheral blood and sputum of patients treated with or or without benralizumab. Determination of IL5Rα levels will be performed by flow cytometry

DETAILED DESCRIPTION:
For this:

1. Investigators will monitor basophil miRNAs changes with benralizumab analyzing miRNAS profile of isolated basophil before and after benralizumab treatment.
2. Also, in vitro characterization of benralizumab effects on functionality of human basophils (isolated from allergic asthmatic patients) and human cell line KU812, measuring apoptosis, activation, degranulation and histamine release will be performed.

ELIGIBILITY:
Inclusion Criteria:

* .It is mandatory that all patients can comprehend the study requirements and provide informed consent for their participation in MEGA.

Group A:

* Adult people (≥ 18 and ≤ 80 years old) with eosinophilic severe asthma requiring high-dose inhaled corticosteroids plus long-acting beta agonists (with or without long-acting muscarinic antagonist or Montelukast or oral corticosteroids)
* Benralizumab treatment approved.

Group B:

.Patients with allergic asthma (prick test or RAST positive).

Exclusion Criteria:

* Patients with continuous OCS treatment
* Patients with Immunosuppressive drugs
* Patients with primary or secondary immune deficiency,
* Patients with chronic or/and concomitant disease, presence of severe systemic disease or cancer,
* Patients with possible infestation by parasites.
* Patients with other acute or chronic active lung disorders Patients with significant psychiatric disorders
* Patients with biological treatment will be excludes for group B

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Group A: f patients with severe eosinophilic uncontrolled asthma treated with Benralizumab Those will be patients with severe eosinophilic asthma who are being treated with benralizumab and who want to participate in a volunteer manner in the study after signing informed consent. The decision of the patients treatment with benralizumab included in the study will not come in any case influenced by their participation in the study but will be made in accordance with the clinical criteria established by the Asthma Multidisciplinary Unit (UMA).
  Group B:patients with allergic asthma without indication of treatment with biological therapy.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Fold changes in number of basophils | From 1 to 12 months
  Fold changes in number of basophils after 8 week, 6 months and 1 year of benralizumab treatment (Fasenra®, Astra Zeneca) in blood and sputum in patients with severe eosinophilic asthma
Fold changes in number of innate inmmune cells | From 1 to 12 months
  Fold changes in number of innate immune cells s after 8 week, 6 months and 1 year of benralizumab treatment (Fasenra®, Astra Zeneca) in blood and sputum in patients with severe eosinophilic asthma
The fold changes of IL-5R expression in basophils | From 1 to 12 months
  The fold changes of IL-5R expression in basophils after 8 week, 6 months and 1 year of benralizumab treatmen
The fold changes of f IL-5R expression in innate lymphoid cells | From 1 to 12 months
  The fold changes of f IL-5R expression in innate lymphoid cells after 8 week, 6 months and 1 year of benralizumab treatment

SECONDARY OUTCOMES:
Fold changes of miRNAs profile in basophils | From 6 to 18
  1. Fold changes of miRNAs profile in basophils after tratment of Benralizumab in in patients with severe eosinophilic asthma treatment.
Fold changes of serum IL-5R | Fromm 6 to 12
  Fold changes of serum IL-5R (microg/ml) in patients treated with benralizumab
Effect of benralizumab in basophil apoptosis | From 12 to 24 months
  The effect of benralizumab in basophil apoptosis isolated from from allergic asthmatic patients will be measure by fold change of annexin V
Effect of benralizumab in KU812 apoptosis | From 12 to 24 months
  The effect of benralizumab in KU812 apoptosis will be measure by fold change of annexin V in KU812 cultures
Effect of benralizumab in basophil activation | From 12 to 24 months
  The effect of benralizumab in basophil activation isolated from from allergic asthmatic patients will be measur by fold change of CD63, and CD203C on membrane by flow cytometry
Effect of benralizumab in KU812 activation | From 12 to 24 months
  The effect of benralizumab in KU812 activation will be measurie by fold change of CD63, and CD203C on membrane by flow cytometry
Effect of benralizumab in basophil degranulation | From 12 to 24 months
  The effect of benralizumab in basophil degranulation will be measure by histamine releasing in isolated basophils from from allergic asthmatic patients
Effect of benralizumab in KU812 degranulation | From 12 to 24 months
  The effect of benralizumab in basophil degranulation will be measure by histamine releasing in KU812 cultured cells

CONTACTS AND LOCATIONS:
Overall Officials: VICTORIA DEL POZO, PhD, Principal Investigator — IIS-FUNDACIÓN JIMENEZ DIAZ
Locations (1):
- Instituto Investigación FJD, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided